CLINICAL TRIAL: NCT05271890
Title: Rheumatoid Arthritis and Treatment of Periodontitis: a Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Filippo Graziani, DDS MClinDent PhD, FULL PROFESSOR, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Perioreuma
Record Dates: First submitted 2022-02-27; First posted 2022-03-09 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Periodontitis; Arthritis, Rheumatoid
Keywords: Periodontitis; Rheumatoid arthritis; Treatment of periodontitis
MeSH Terms: conditions — Periodontitis; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate periodontal treatment (Experimental): Subjects assigned to this group were receiving non-surgical periodontal treatment as well as oral hygiene instructions immediately after their inclusion. All subjects were undergone full periodontal and rheumatologic clinical examinations both at baseline and 90 days after the completion of the treatment. Blood collection for the analysis of the serum concentration of CRP, ESR, Fibrinogen, IL-6 and TNF-α was also performed at baseline and 90 days after periodontal treatment.
  Interventions: Procedure: Immediate non-surgical periodontal treatment and oral hygiene instructions
- Delayed periodontal treatment (No Intervention): Subjects assigned to this group were receiving non-surgical periodontal treatment 90 days after baseline evaluation. All subjects were undergone full periodontal and rheumatologic clinical examinations both at baseline and 90 days after. Blood collection for the analysis of the serum concentration of CRP, ESR, Fibrinogen, IL-6 and TNF-α was also performed at baseline and 90 days after.

INTERVENTIONS:
Procedure: Immediate non-surgical periodontal treatment and oral hygiene instructions
  Arms: Immediate periodontal treatment

SUMMARY:
Periodontitis is an infectious disease defined by bacteria-mediated inflammation of the supporting tissues of the teeth that if left untreated may ultimately lead to the destruction of the attachment apparatus, culminating in tooth loss. Rheumatoid arthritis is a chronic destructive inflammatory disease characterized by autoantibodies and the accumulation and persistence of an inflammatory infiltrate in the synovial membrane that leads to synovitis and the destruction of the joint architecture. The objective of this study was to evaluate the possible beneficial additional value of non-surgical periodontal therapy on systemic markers of inflammation and clinical and serological parameters of rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects affected by rheumatoid arthritis with a stable therapeutic regimen for at least 3 months preceding the study participation
* Subjects with at least 15 teeth
* Subjects affected by severe generalized periodontitis that had undergone no periodontal treatment in the 6 months preceding the study participation

Exclusion Criteria:

* Age younger than 18 years
* Pregnancy or breastfeeding
* Edentulism
* Diagnosis of other autoimmune pathologies, liver disease, diabetes, early/juvenile arthritis or syndromes associated with RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08-25 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Disease Activity Score 28 (DAS-28) | 90 days
  Variation of DAS-28 90 days after periodontal treatment

SECONDARY OUTCOMES:
Erythrocyte Sedimentation Rate (ESR) | 90 days
  Variation of ESR 90 days after periodontal treatment
C-Reactive Protein (CRP) | 90 days
  Variation of CRP 90 days after periodontal treatment
Interleuchin-6 concentration (IL-6) | 90 days
  Variation of IL-6 90 days after periodontal treatment
Oral Health Related Quality of Life (OHRQoL) | 90 days
  Variation of OHRQoL 90 days after periodontal treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pisa, Pisa, Italy